CLINICAL TRIAL: NCT03956550
Title: A Randomized, Double-Blind, Multi-Dose, Placebo-Controlled Study to Evaluate the Efficacy and Safety of REGN5069 in Patients With Pain Due to Osteoarthritis of the Knee
Brief Title: A Study to Examine the Efficacy and Safety of REGN5069 in Patients With Pain Due to Osteoarthritis of the Knee
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Regeneron has discontinued further clinical development of REGN5069, an antibody to GFRα3, which was previously being studied in osteoarthritis pain of the knee
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R5069-OA-1849
Record Dates: First submitted 2019-05-16; First posted 2019-05-20 (Actual); Results first posted 2021-07-01 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Osteoarthritis of the Knee; Pain
MeSH Terms: conditions — Osteoarthritis, Knee; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- REGN5069 Low Dose (Experimental): Randomized in a 1:1:1 ratio
  Interventions: Drug: REGN5069
- REGN5069 High Dose (Experimental): Randomized in a 1:1:1 ratio
  Interventions: Drug: REGN5069
- Matching Placebo (Experimental): Randomized in a 1:1:1 ratio
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: REGN5069 — Intravenous (IV) Dose every 4 weeks (Q4W)
  Arms: REGN5069 High Dose; REGN5069 Low Dose
Drug: Matching Placebo — Intravenous (IV) Dose every 4 weeks (QW4)
  Arms: Matching Placebo

SUMMARY:
The primary objective of the study is to evaluate the efficacy of REGN5069 compared to placebo in patients with pain due to radiographically-confirmed OA of the knee who have a history of inadequate joint pain relief or intolerance to current analgesic therapy.

The secondary objectives of the study are:

* To characterize the concentrations of functional REGN5069 in serum over time when patients are treated for up to 12 weeks
* To assess the safety and tolerability of REGN5069 compared with placebo when patients are treated for up to 12 weeks
* To measure levels of anti-drug antibodies (ADAs) against REGN5069 following multiple IV administrations

ELIGIBILITY:
Key Inclusion Criteria:

* Generally in good health at the screening visit
* Body mass index (BMI) ≤39 kg/m2 at the screening visit
* Clinical diagnosis of OA of the knee on the American College of Rheumatology criteria (Altman, 1986) with radiologic evidence of OA (K-L score ≥2) at the index joint at the screening visit
* Moderate-to-severe pain in the index joint
* A history of inadequate pain relief from or intolerance to analgesics used for OA

Key Exclusion Criteria:

* Diagnosis of systemic diseases that may affect joints
* History or presence of osteonecrosis, destructive arthropathy, neuropathic joint arthropathy, pathologic fractures in any shoulder, hip, or knee joint(s), hip dislocation (prosthetic hip dislocation is eligible), or knee dislocation (patella dislocation is eligible) at the screening visit. Presence of subchondral insufficiency fracture on screening films or MRI as assessed by the central imaging reader.
* Is scheduled for a joint replacement surgery to be performed during the study period
* Received an intra-articular injection of hyaluronic acid in any joint within 90 days prior to the screening visit
* Systemic (ie, IV, oral, or intramuscular) corticosteroids within 30 days prior to the screening visit. Intra-articular corticosteroids in the index joint within 12 weeks prior to the screening visit, or to any other joint within 30 days prior to the screening visit (topical, intranasal, or inhaled corticosteroids are permitted).
* History or presence at the screening visit of multiple sclerosis, autonomic neuropathy, diabetic neuropathy, or other peripheral neuropathy
* Significant concomitant illness including, but not limited to, psychiatric, cardiac, renal, hepatic, neurological, endocrinological, metabolic, or lymphatic disease that, in the opinion of the investigator, would adversely affect the patient's participation in the study
* History of myocardial infarction, acute coronary syndromes, transient ischemic attack, or cerebrovascular accident within 12 months prior to the screening visit

Note: Other protocol defined inclusion/exclusion criteria apply.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 259 (Actual)
Dates: Start 2019-05-21 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-10-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (12):
- United States (4):
  - Regeneron Study Site, DeLand, Florida
  - Regeneron Study Site, Jupiter, Florida
  - Regeneron Study Site, Miami, Florida
  - Regeneron Study Site, Charleston, South Carolina
- Regeneron Study Site, Tbilisi, Georgia
- Regeneron Study Site, Chisinau, Moldova
- Poland (5):
  - Regeneron Study Site, Lublin, Lublin Voivodeship
  - Regeneron Study Site, Zamość, Lublin Voivodeship
  - Regeneron Study Site, Warsaw, Masovian Voivodeship
  - Regeneron Study Site, Bialystok, Podlaskie Voivodeship
  - Regeneron Study Site, Zgierz, Łódź Voivodeship
- Regeneron Study Site, Kyiv, Ukraine

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Individual anonymized participant data will be considered for sharing once the indication has been approved by a regulatory body, if there is legal authority to share the data and there is not a reasonable likelihood of participant re-identification.
Access Criteria: Qualified researchers may request access to anonymized patient level data or aggregate study data when Regeneron has received marketing authorization from major health authorities (e.g., FDA, EMA, PMDA, etc) for the product and indication, has the legal authority to share the data, and has made the study results publicly available (eg, scientific publication, scientific conference, clinical trial registry).
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 5 countries and 12 sites participated in enrollment. It consisted of screening period up to 30 days, followed by a 12-week randomized, double-blind, placebo-controlled treatment period, a 24-week follow-up period, and end-of-study phone call approximately 52 weeks after first dose. Study was terminated after all participants completed the week 36 visits.
Pre-assignment Details: A total of 259 participants were randomized in 1:1:1 ratio to receive REGN5069 at 100 mg IV Q4W, REGN5069 at 1000 mg IV Q4W, or matching placebo Q4W. Participants were to receive 3 fixed-dose IV infusions at baseline, week 4, and week 8. 171 participants were randomized to receive REGN5069 (86 participants in the 100 mg Q4W group and 85 in the 1000 mg Q4W group) and 88 were randomized to receive placebo.
Groups:
- Placebo: Participants received matching placebo intravenously every 4 weeks (Q4W)
- REGN5069 100 mg Q4W: Participants received 100 milligrams (mg) of REGN5069 intravenously every 4 weeks (Q4W)
- REGN5069 1000 mg Q4W: Participants received 1000 milligrams (mg) of REGN5069 intravenously every 4 weeks (Q4W)
Period: Overall Study
Arm/Group | Placebo | REGN5069 100 mg Q4W | REGN5069 1000 mg Q4W
Started | 88 | 86 | 85
Completed | 18 | 14 | 15
Not Completed | 70 | 72 | 70
Not completed — Sponsor decision | 65 | 66 | 64
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Withdrawal by Subject | 5 | 5 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | REGN5069 100 mg Q4W | REGN5069 1000 mg Q4W | Total
Number analyzed (Participants) | 88 | 86 | 85 | 259
Age, Continuous [Mean (Standard Deviation); unit: Years] — Full analysis set population (FAS): included all randomized participants
  Years | 63.5 (8.27) | 63.9 (7.39) | 64.7 (8.30) | 64.0 (7.98)
Sex: Female, Male [Count of Participants; unit: Participants] — Full analysis set population (FAS): included all randomized participants
  Participants
    Female | 64 | 74 | 68 | 206
    Male | 24 | 12 | 17 | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Full analysis set population (FAS): included all randomized participants
  Participants
    Hispanic or Latino | 4 | 1 | 2 | 7
    Not Hispanic or Latino | 84 | 85 | 83 | 252
    Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants] — Full analysis set population (FAS): included all randomized participants
  Participants
    White | 83 | 85 | 81 | 249
    Black or African American | 5 | 1 | 4 | 10
    Asian | 0 | 0 | 0 | 0
    American Indian or Alaska Native | 0 | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Not reported | 0 | 0 | 0 | 0
    Other | 0 | 0 | 0 | 0
Western Ontario and McMaster Osteoarthritis Index (WOMAC) Pain Subscale Score [Mean (Standard Deviation); unit: Scores on a scale] — The WOMAC index is comprised of 24 parameters grouped in 3 subscales (pain-5 questions, physical function -17 questions and stiffness - 2 questions), with 0-10 grading of each question. The scores for each subscale are summed up, divided by number of questions, and each subscale is reported using Numerical Rating Scale score of 0-10. In addition to subscales, a total score is provided as the sum of normalized subscale scores divided by three, and reported using a Numerical Rating Scale score of 0-10. Higher scores indicate worse pain, stiffness and functional limitations. Population: Here 'n' = number of evaluable participants at this time interval
  Scores on a scale
    number analyzed (Participants) | 87 | 86 | 85 | 258
    (all) | 6.68 (1.257) | 6.24 (1.203) | 6.47 (1.150) | 6.36 (1.179)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 12 in the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Score
Description: The WOMAC index is comprised of 24 parameters grouped in 3 subscales (pain-5 questions, physical function -17 questions and stiffness - 2 questions), with 0-10 grading of each question. The scores for each subscale are summed up, divided by number of questions, and each subscale is reported using Numerical Rating Scale score of 0-10. In addition to subscales, a total score is provided as the sum of normalized subscale scores divided by three, and reported using a Numerical Rating Scale score of 0-10. Higher scores indicate worse pain, stiffness and functional limitations.
Time Frame: Baseline to Week 12
Population: Full analysis set population (FAS): included all randomized participants; Here 'n' = number of evaluable participants at the specific time point.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | REGN5069 100 mg Q4W | REGN5069 1000 mg Q4W
Number analyzed (Participants) | 84 | 80 | 82
Scores on a scale | -2.09 (0.188) | -2.37 (0.191) | -1.98 (0.190)
Statistical Analysis 1: Comparison: Placebo vs REGN5069 100 mg Q4W; Test type: Superiority; p = 0.2978, Mixed Models Analysis
Statistical Analysis 2: Comparison: Placebo vs REGN5069 1000 mg Q4W; Test type: Superiority; p = 0.6890, Mixed Models Analysis

2. Secondary Outcome: Change From Baseline to Week 12 in WOMAC Total Score
Description: as for outcome 1
Time Frame: Week 12
Population: Full analysis set population (FAS): included all randomized participants; Here "number analyzed" = number of evaluable participants at this time interval
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | REGN5069 100 mg Q4W | REGN5069 1000 mg Q4W
Number analyzed (Participants) | 84 | 80 | 82
Scores on a scale | -1.83 (0.177) | -2.15 (0.179) | -1.81 (0.181)
Statistical Analysis 1: Comparison: Placebo vs REGN5069 100 mg Q4W; Test type: Superiority; p = 0.1973, Mixed Models Analysis
Statistical Analysis 2: Comparison: Placebo vs REGN5069 1000 mg Q4W; Test type: Superiority; p = 0.9420, Mixed Models Analysis

3. Secondary Outcome: Change From Baseline to Week 12 in WOMAC Physical Function Subscale Score
Description: as for outcome 1
Time Frame: Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | REGN5069 100 mg Q4W | REGN5069 1000 mg Q4W
Number analyzed (Participants) | 84 | 80 | 82
Scores on a scale | -1.74 (0.180) | -2.09 (0.183) | -1.75 (0.182)
Statistical Analysis 1: Comparison: Placebo vs REGN5069 100 mg Q4W; Test type: Superiority; p = 0.1597, Mixed Models Analysis
Statistical Analysis 2: Comparison: Placebo vs REGN5069 1000 mg Q4W; Test type: Superiority; p = 0.9719, Mixed Models Analysis

4. Secondary Outcome: Change From Baseline to Week 12 in Patient Global Assessment (PGA) Score
Description: The Patient Global Assessment of OA (PGA) is a patient-rated assessment of current disease state on a 5-point Likert scale (1 = very good; 2 = good; 3 = fair; 4 = poor; and 5 = very poor).
Time Frame: Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | REGN5069 100 mg Q4W | REGN5069 1000 mg Q4W
Number analyzed (Participants) | 84 | 80 | 82
Scores on a scale | -0.59 (0.076) | -0.75 (0.078) | -0.80 (0.078)
Statistical Analysis 1: Comparison: Placebo vs REGN5069 100 mg Q4W; Test type: Superiority; p = 0.1365, Mixed Models Analysis
Statistical Analysis 2: Comparison: Placebo vs REGN5069 1000 mg Q4W; Test type: Superiority; p = 0.0604, Mixed Models Analysis

5. Secondary Outcome: Change From Baseline to Week 12 in WOMAC Stiffness Subscale Score
Description: as for outcome 1
Time Frame: Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | REGN5069 100 mg Q4W | REGN5069 1000 mg Q4W
Number analyzed (Participants) | 84 | 80 | 82
Scores on a scale | -1.70 (0.214) | -2.20 (0.217) | -1.88 (0.217)
Statistical Analysis 1: Comparison: Placebo vs REGN5069 100 mg Q4W; Test type: Superiority; p = 0.0989, Mixed Models Analysis
Statistical Analysis 2: Comparison: Placebo vs REGN5069 1000 mg Q4W; Test type: Superiority; p = 0.5487, Mixed Models Analysis

6. Secondary Outcome: Percentage of Participants With ≥30% Improvement in WOMAC Pain Subscale Score
Description: as for outcome 1
Time Frame: Week 12
Population: Full analysis set population (FAS): included all randomized participants
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | REGN5069 100 mg Q4W | REGN5069 1000 mg Q4W
Number analyzed (Participants) | 88 | 86 | 85
Percentage of participants | 51.1 | 58.1 | 47.1
Statistical Analysis 1: Comparison: Placebo vs REGN5069 100 mg Q4W; Test type: Superiority; p = 0.3572, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo vs REGN5069 1000 mg Q4W; Test type: Superiority; p = 0.5747, Cochran-Mantel-Haenszel

7. Secondary Outcome: Number of Non-Serious and Serious Treatment-Emergent Adverse Events (TEAEs) Through End of Study
Description: An adverse event (AE) is any untoward medical occurrence in a patient administered a study drug which may or may not have a causal relationship with the study drug. Treatment-emergent AEs (TEAEs) are AEs that developed or worsened during the treatment period.
Time Frame: Baseline to Week 36
Population: Safety Analysis Set (SAF): included all randomized participants who received any study drug
Measure: Number; unit: Events
Arm/Group | Placebo | REGN5069 100 mg Q4W | REGN5069 1000 mg Q4W
Number analyzed (Participants) | 88 | 85 | 84
Events
  Non-Serious TEAEs | 78 | 42 | 55
  Serious TEAEs | 0 | 2 | 0

8. Secondary Outcome: Number of Imaging Abnormalities Consistent With Adjudicated Arthropathies Through End of Study
Description: Adjudicated arthropathy is an umbrella term referring to Rapidly Progressive Osteoarthritis Type 1 (RPOA-1), Rapidly Progressive Osteoarthritis Type 2 (RPOA-2), subchondral insufficiency fractures (SIF) and osteonecrosis (ON) confirmed by an arthropathy adjudication committee.
Time Frame: Baseline to Week 36
Population: Safety Analysis Set (SAF): included all randomized participants who received any study drug
Measure: Number; unit: Events
Arm/Group | Placebo | REGN5069 100 mg Q4W | REGN5069 1000 mg Q4W
Number analyzed (Participants) | 88 | 85 | 84
Events
  Baseline Up to and Including Week 12 Visit | 1 | 0 | 0
  After Week 12 Visit, Up to and Including Week 36 | 0 | 0 | 0

9. Secondary Outcome: Number of Participants With Presence of Anti-REGN5049 Antibody Development Through End of Study
Description: Immunogenicity will be characterized by ADA responses & titers. Responses categories: Negative - ADA negative response at all time points, regardless of missing samples; Pre-existing immunoreactivity - ADA positive response at baseline with all post first dose negative results or positive response at baseline with all post first dose ADA responses < 9-fold over baseline titer levels; Treatment-boosted response - positive response in the assay post first dose, ≥ 9-fold over baseline titer levels, when baseline results are positive; Treatment-emergent response - ADA positive response in the REG5069 ADA assay post first dose when baseline results = negative or missing.
Time Frame: Baseline to Week 36
Population: Anti-Drug Antibody (ADA) Analysis Set: included all treated participants who received any amount of study drug (active or placebo [safety analysis set (SAF)]) and had at least one non-missing anti-REGN5069 antibody result following the first dose of study drug or placebo. ADA analysis set is based on actual treatment received, rather than randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | REGN5069 100 mg Q4W | REGN5069 1000 mg Q4W
Number analyzed (Participants) | 84 | 83 | 82
Participants
  Negative | 82 | 83 | 78
  Pre-Existing Immunoreactivity | 1 | 0 | 4
  Treatment-Boosted Response | 0 | 0 | 0
  Treatment-Emergent Response | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events (AE) and Serious Adverse Events (SAE) were collected from the time of informed consent signature and then at each visit until the end of follow-up visit (week 36) for AEs and until end of study visit (week 52) for SAEs. The study was terminated early at 36 weeks.
Groups:
- REGN5069 100 mg IV Q4W: Participants received 100 milligrams (mg) of REGN5069 intravenously every 4 weeks (Q4W)
- REGN5069 1000 mg IV Q4W: Participants received 1000 milligrams (mg) of REGN5069 intravenously every 4 weeks (Q4W)
Arm/Group | Placebo | REGN5069 100 mg IV Q4W | REGN5069 1000 mg IV Q4W
All-Cause Mortality (participants affected / at risk) | 0/88 | 0/85 | 0/84
Serious Adverse Events (participants affected / at risk) | 3/88 | 3/85 | 0/84
Other Adverse Events (participants affected / at risk) | 48/88 | 33/85 | 36/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=88) | REGN5069 100 mg IV Q4W (N=85) | REGN5069 1000 mg IV Q4W (N=84)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=88) | REGN5069 100 mg IV Q4W (N=85) | REGN5069 1000 mg IV Q4W (N=84)
Headache (Nervous system disorders) | 30 (64) | 19 (36) | 20 (47)
Nasopharyngitis (Infections and infestations) | 11 (14) | 4 (4) | 7 (10)
Urinary tract infection (Infections and infestations) | 9 (14) | 4 (5) | 5 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (14) | 3 (4) | 8 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (7) | 9 (17) | 7 (9)
Toothache (Gastrointestinal disorders) | 10 (15) | 5 (7) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2019-09-04): https://cdn.clinicaltrials.gov/large-docs/50/NCT03956550/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-17): https://cdn.clinicaltrials.gov/large-docs/50/NCT03956550/SAP_001.pdf